CLINICAL TRIAL: NCT05454462
Title: Double-blind, Vehicle-controlled, Phase I Study to Evaluate Safety and Efficacy of a 0.3% and 1% Topical Formulation of KM-001 for Management of Moderate to Severe Pruritus in Adult Patients With Lichen Simplex Chronicus (LSC)
Brief Title: KM-001 Cream for Treatment of Pruritus in Adult Patients With Lichen Simplex Chronicus (LSC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kamari Pharma Ltd (Network)
Collaborators: Bioskin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KM-001AB1
Record Dates: First submitted 2022-06-29; First posted 2022-07-12 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Lichen Simplex Chronicus
MeSH Terms: conditions — Neurodermatitis | interventions — Hematologic Tests; Urinalysis; Electrocardiography; Pregnancy Tests; Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Topical application of approximately 1 g cream per defined treatment area (2% body surface area [BSA] including target lesion [minimum 0.5% to maximum 2% BSA]) twice daily during a 4-week treatment period (on Days 0 to 27 and one additional application in the morning of Day 28, i.e., 57 treatments)
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be performed double-blind. Double-blind means that neither the patient nor the investigational staff (investigator, study nurse, evaluators, etc.) will know which IMP a patient is receiving.
  This is to ensure that the evaluations are carried out without bias. The IMPs will be blinded by the manufacturer via the labelling procedure. IMPs will be identical in appearance and will be packaged identically so that treatment blind is maintained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KM-001 0.3% (Experimental): KM-001 0.3% cream will be applied to the affected area twice daily for 4 consecutive weeks.
  Interventions: Drug: IMP Application KM-001; Diagnostic Test: Chemistry; Diagnostic Test: Hematology; Diagnostic Test: Urinalysis; Diagnostic Test: Serelogy; Diagnostic Test: 12-Lead ECG; Diagnostic Test: Pregnancy test; Diagnostic Test: Blood PK sampling; Procedure: Physical Examination; Procedure: Vital signa; Diagnostic Test: Investigator's Global Assessment; Diagnostic Test: Itch Assessment via PP-NRSj; Other: E-diary data
- KM-001 1% (Experimental): KM-001 0.3% cream will be applied to the affected area twice daily for 4 consecutive weeks.
  Interventions: Drug: IMP Application KM-001; Diagnostic Test: Chemistry; Diagnostic Test: Hematology; Diagnostic Test: Urinalysis; Diagnostic Test: Serelogy; Diagnostic Test: 12-Lead ECG; Diagnostic Test: Pregnancy test; Diagnostic Test: Blood PK sampling; Procedure: Physical Examination; Procedure: Vital signa; Diagnostic Test: Investigator's Global Assessment; Diagnostic Test: Itch Assessment via PP-NRSj; Other: E-diary data
- Vehicle arm (Placebo Comparator): Vehicle cream will be applied to the affected area twice daily for 4 consecutive weeks.
  Interventions: Drug: IMP Application KM-001; Diagnostic Test: Chemistry; Diagnostic Test: Hematology; Diagnostic Test: Urinalysis; Diagnostic Test: Serelogy; Diagnostic Test: 12-Lead ECG; Diagnostic Test: Pregnancy test; Diagnostic Test: Blood PK sampling; Procedure: Physical Examination; Procedure: Vital signa; Diagnostic Test: Investigator's Global Assessment; Diagnostic Test: Itch Assessment via PP-NRSj; Other: E-diary data

INTERVENTIONS:
Drug: IMP Application KM-001 — KM-001 will be supplied in glass jars (30 ml) and will be provided to patients with spatulas and polyethylene gloves on all the clinical visits. the patient will use IMP twice a day for 28 days.
  Other Names: Experimental drug administration
Diagnostic Test: Chemistry — patients will provide a blood sample for a chemistry blood test on days -14 (screening visit), Day 7(visit 3), day 28 (end of treatment) or at ET visit.
  Other Names: Blood test
Diagnostic Test: Hematology — patients will provide a blood sample for a hematology blood test on days -14 (screening visit), Day 7(visit 3), day 28 (end of treatment) or at ET visit.
  Other Names: Blood test
Diagnostic Test: Urinalysis — Patients will provide a blood sample for a urine test on days -14 (screening visit), Day 7(visit 3), day 28 (end of treatment) or at ET visit.
  Other Names: Urine test
Diagnostic Test: Serelogy — Patients will provide a blood sample for serelogy test at day -14 (screening visit)
  Other Names: Blood test
Diagnostic Test: 12-Lead ECG — patients will undergo an ECG examination on days -14 (screening visit), and day 28 (end of treatment visit).
Diagnostic Test: Pregnancy test — Women of child-bearing potential only will provide at all the on-site visits b-hCG concentration will be tested
  Other Names: Blood test
Diagnostic Test: Blood PK sampling — PK test will be performed on day 1, 7, 28, 35 and on ET visit
Procedure: Physical Examination — patients will undergo a physical examination on all the clinical visits
Procedure: Vital signa — patient's vital signs will be measured on all the clinical visits
Diagnostic Test: Investigator's Global Assessment — patient's disease evaluations will be evaluated on all the clinical visits
  Other Names: score
Diagnostic Test: Itch Assessment via PP-NRSj — patient's disease evaluations will be evaluated on all the clinical visits
  Other Names: score
Other: E-diary data — The patient will record IMP adminidsration and AE events in a diary every day throughout the all study period

SUMMARY:
This is a phase 1, multi-center, randomized, vehicle-controlled, double-blinded, parallel-group study.

Approximately 6 sites will conduct the study at Germany. Approximately 61 patients (male and female) planned to be screened. 51 patient planned to be randomized.

Patients will be randomized to 1 of 3 treatment arms (KM-001 0.3%, KM-001 1%, or vehicle cream) iina a ration of 1:1:1

Patient's duration of participation will be up to 7 weeks,

* a screening period with 1 visit (Visit 1) within up to 14 days (Days -14 to -1),
* a 4-week treatment period with 3 visits (Visit 2 on Day 0, Visit 3 on Day 7, Visit 4 at Day 28 and 2 phone calls on Days 14 and 21, and
* a 1-week follow-up period with 1 visit (Visit 5 on Day 35), as well as unscheduled visits as needed

Since KM-001 is tested in humans for the first time, the safety of KM-001 will be evaluated in a subgroup of 6 patients (sentinel group) at selected sites prior to screening of the remaining sites.

Efficacy assessments will include subjective assessments of itch and investigator assessment of the treatment effect on LSC target lesion using scoring systems.

Safety parameter (including physical examination, vital signs, ECG, standard laboratory test, and PK analysis) will be monitored from the signing of the informed consent form (ICF) until the last follow-up visit. Recording of AEs and serious AEs (SAEs) will be done throughout the study with special attention to local AEs in the treatment area (LSC target lesion, dermal safety).

DETAILED DESCRIPTION:
This phase I study will be performed in patients with LSC instead of healthy subjects as in these patients, the significant histological changes (acanthosis and parakeratosis) result in heavily altered physiology and anatomy of the skin and any data including tolerability generated by administering the IMP on healthy skin can hardly be extrapolated to patients with LSC.

The setting can be compared with early studies in Psoriasis patients where it is established to include patients from the beginning. Based on preclinical experiments, no pharmacological relevant systemic absorption is expected.

PK sampling will be done for confirmation. Parallel group comparison is a common method and provides optimal conditions for examining efficacy. Comparisons to a vehicle is a common procedure. Randomization provides the most reliable and impartial method of determining differences between treatments as in this case active versus vehicle.

Double-blind conditions minimize any possible observer bias regarding treatment effects.

A vehicle control is included to evaluate the efficacy, safety, and tolerability of the cream without the active ingredient and to differentiate whether the drug substance or the drug product might cause any effects.

A duration of a 4-week treatment period is assumed to be appropriate to assess efficacy, safety, and tolerability based on preclinical data

ELIGIBILITY:
Inclusion Criteria:

1. Read, understood, and signed an ICF before any investigational procedure(s) are performed.
2. Male or female and aged ≥18 to 75 years at the time of screening.
3. Chronic moderate to severe pruritus defined as:

   1. Itching that has been present for 6 weeks or more prior to the screening AND
   2. At the screening visit (Visit 1) and enrollment visit (Visit 2): peak pruritus-numerical rating scale (PP-NRS)24h is ≥7.
4. Clinical diagnosis of LSC for at least 8 weeks prior to screening:

   1. LSC lesions defined as dry, scaly, thickened plaques of skin (lichenification) caused by repeated rubbing or scratching, on upper limbs, trunk, and/or lower limbs.
   2. To have no more than 3 lesions, total size not exceeding 5% of BSA from which one (target lesion) will be selected for treatment (minimum area of lesion selected for treatment: 0.5% BSA).
5. Female patients of childbearing potential1 must use a highly effective birth control method(failure rate ˂1% per year when used consistently and correctly) (17) throughout the study and for at least 4 weeks after last application of IMP.

In addition to the hormonal contraception, female patients must agree to use a supplemental barrier method during intercourse with a male partner (i.e., male condom) throughout the study and for at least 4 weeks after last application of IMP.

Female patients must be having regular menstrual periods (interval of 21-35 days, duration of 2-7 days for several months) at the baseline visit (as reported by the patient); exception: patients using hormonal contraceptives that preclude regular menstrual periods, menopausal or hysterectomized patients. A male patient with a pregnant or non-pregnant female partner of childbearing potentialmust use adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice; as a minimum, the male patient must agree to use condom during treatment and until the end of relevant systemic exposure in the male subject (7 days post-treatment).

Male patients must refrain from sperm donation throughout the study and for 7 days after the last study drug administration.

7. Female patients of non-childbearing potential must meet one of the following criteria:

1. Absence of menstrual bleeding for 1 year prior to screening without any other medical reason.
2. Documented hysterectomy or bilateral oophorectomy at least 3 months before the study.

   8. Patient is willing and able to comply with all of the time commitments and procedural requirements of this CTP, including daily e-diary recordings by the patient using an electronic handheld device and an internet connection during the study.

Exclusion Criteria:

1. Known hypersensitivity or any suspected cross-allergy to the active pharmaceutical ingredient (API) and/or excipients.
2. Chronic pruritus resulting from another active condition other than LSC such as, but not limited to, psoriasis, atopic dermatitis, lichen planus contact dermatitis, folliculitis, habitual picking, bullous autoimmune disease, neuropathy.
3. Genital, anal or scalp LSC.
4. History of or current confounding skin condition (psoriasis, cutaneous T-cell lymphoma [mycosis fungoides or Sezary syndrome], chronic actinic dermatitis with [present or previous] skin cancer on the site of LSC, bullous disorders, dermatitis herpetiformis).
5. Cutaneous infection within 1 week before the screening visit or any infection requiring treatment with oral, parenteral antibiotics, antivirals, antiparasitics or antifungals or any topical within 1 week before the screening visit. Patients may be rescreened once the infection has resolved.
6. Positive hepatitis B surface antigen [HBsAg], hepatitis B core antibody [HBcAb], hepatitis C antibody, or human immunodeficiency virus antibody serology results at the screening visit.
7. Patients with active atopic dermatitis.
8. Neuropathic and psychogenic pruritus, such as, but not limited to, notalgia paresthetica, brachioradial pruritus, small fiber neuropathy, skin picking syndrome, or delusional parasitosis.
9. Patients with the following medical conditions:

   1. High blood pressure (BP), defined as resting systolic BP ≥140 mmHg and/or diastolic BP ≥90 mmHg (according to 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice [18]).
   2. Patients with poorly controlled and/or complicated (retinopathy/nephropathy/neuropathy) diabetes glycosylated hemoglobin (HbA1c) of >7%, fasting serum glucose >130 mg/dl.
   3. Patients with history of angina pectoris and/or myocardial infarction.
   4. Systemic autoimmune conditions (including, but NOT limited to: systemic lupus erythematosus, rheumatoid arthritis etc.).
   5. Small fiber neuropathy.
   6. Any other condition that could, in the investigator's opinion, affect patient safety, his ability to participate in the study or ability of the investigator to assess the skin.
10. Having received any of the prohiboted treatments in Table 1 within the specified timeframe before the baseline visit.
11. Pregnant women (positive serum pregnancy test result at the screening and baseline visits), breastfeeding women, or women planning a pregnancy during the clinical trial.
12. History of lymphoproliferative disease or history of malignancy of any organ system within the last 5 years, except for:

    1. Basal cell carcinoma, squamous cell carcinoma in situ (Bowen's disease), or carcinomas in situ of the cervix that had been treated and with no evidence of recurrence in the last 52 weeks before the baseline visit, or;
    2. Actinic keratoses that had been treated and with no evidence of recurrence in the last 8 weeks.
13. Any known or suspected state of immunodeficiency due to primary or secondary immunodeficiency syndromes, organ transplants (except corneal transplant), previous opportunistic infection, or any other state of immunodeficiency as judged by the investigator.
14. Any clinically relevant disorder or abnormal finding which could affect the safety of the patient throughout the study and/or impede the patient's ability to complete the study, as assessed by the investigator.
15. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or bilirubin exceeding the upper limit of normal (ULN), or any other laboratory abnormalities considered clinically relevant by the investigator, at the screening/baseline visit.
16. Any condition that may put the patient at significant risk according to the investigator's judgment.
17. Any disorder which may interfere with study assessments (e.g., poor venous access or needle-phobia).
18. Major surgical procedure planned or expected during the clinical trial.
19. Patient is unwilling to refrain from using prohibited medications during the clinical trial.
20. Currently participating or participated in any other study of a drug or device, within the past 2 months before the screening visit, or is in an exclusion period (if verifiable) from a previous study.
21. Close affiliation with the investigator (e.g., a close relative) or persons working at bioskin GmbH or the study sites or patient is an employee of sponsor.
22. Patient is institutionalized because of legal or regulatory order.
23. Patients who have been administered any vaccine for COVID-19 within 30 days prior to first treatment.
24. Tattoos and scars in the areas to be treated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Safety endpoint - Will be assessed through collection and analysis of adverse events | up to 7 weeks
  Incidence of treatment-emergent adverse events (AEs) and serious adverse events (SAEs)
Safety endpoint-Hematology blood test | up to 7 weeks
  RBC, WBC and platelets count, absolute neutrophils, lymphocytes, monocytes, eosinophil and basophil counts, reticulocyte count, hemoglobin, hematocrit, MCV and MCH will be tested and assess.
  The assessment will be compared thr baseline results. Exceptional values above the normal or below the normal will indicate an aggravation of the participant's condition
Safety endpoint- Serology blood test - HBV | up to 14 days
  HBsAb,HBsAg, HBcAb will be prformed at screening visit. laboratory measurements will be assessed and listed.
Safety endpoint- Serology blood test- Hepatits C | up to 14 days
  Hepatits C virus antibody will be prformed at screening visit. laboratory measurements will be assessed and listed.
Safety endpoint- Serology blood test- HIV | up to 14 days
  HIV will be prformed at screening visit. laboratory measurements will be assessed and listed.
Safety endpoint-Chemistry | up to 7 weeks
  Chemistry measurements will be presented descriptively by visit including changes from baseline for quantitative outcomes. Shift tables showing changes with respect to the normal range between baseline and each post-baseline visit will be shown. Incidence of any laboratory outcome of clinical significance will be shown for scheduled and unscheduled measures, including a presentation for each laboratory parameter.
Safety endpoin-Urine tests | up to 7 weeks
  Specific gravity, pH, glucose, protein, blood and ketones by will perform by dipstick. assessment will be compared to the normal range.
  Change from baseline (Day -14 to -1 [screening/Visit 1]) in safety laboratory parameters at Day 7 (Visit 3 or ETV) and Day 28 (Visit 4 or ETV)
Safety endpoin-Pregnancy test | up to 7 weeks
  In women of child-bearing potential only. At all the on-site visits serum beta-human chorionic gonadotropin (b-hCG) concentration will be tested.
Safety endpoin-Vital signs- Pulse | up to 7 weeks
  units: BPM (beats per minute) Data management team will assess and review the vital signs. The category of the assessments will be compared to the normal ranges. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition
Safety endpoin-Vital signs- Blood pressure | up to 7 weeks
  units: blood pressure [mm Hg]. Data management team will assess and review the vital signs. The category of the assessments will be compared to the normal ranges. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition
Safety endpoin-Vital signs- Body temperature | up to 7 weeks
  body temperature will be assesed and the changes from the baseline. units:Celsius degrees. Data management team will assess and review the vital signs. The category of the assessments will be compared to the normal ranges.
Safety endpoin-Electrocardiogram | up to 7 weeks
  A 12-lead, resting, digital ECG will be taken for each participant at Screening and on Day 28 or at ETV. the following ECG parameters will be recorded: heart rate (HR), PR, QT and QRS intervals and QTC. Resting ECG parameter and changes from baseline will be assesed
Safety endpoin-Physical examination | up to 4 weeks
  A complete examination will be performed at screening and baseline: As a minimum, the following body systems will be examined and listed: basic status of the main organ systems (ear nose throat, heart, lungs, abdomen, neurological status) as well as physical examination of the skin.
  An abbreviated examination including a comprehensive skin examination will be performed at other indicated visits.
  Height and weight measurement will be performed at screening only.
KM-001 plasma levels (PK) - Cmax | Up to 5 weeks
  CMAX measurement (mg/ml)
KM-001 plasma levels (PK) - Tmax | Up to 5 weeks
  Tmax measurement (h)
KM-001 plasma levels (PK) - AUC 0-t | Up to 5 weeks
  AUC measurement (mg*h/L)

SECONDARY OUTCOMES:
Efficacy endpoint will be assessed through collection and analysis of lesion Assessment-IGA | up to 7 weeks
  Effect of the treatment on LSC-target lesion, as assessed by location shift in IGA score Effect of the treatment will be assessed using the Investigator's Global Assessment (IGA) scale, which is a 5-point scale (from 0 ="no disease" to 4="severe disease").
Efficacy endpoint will be assessed through collection and analysis of lesion Assessment- (PP-NRS) | up to 7 weeks
  Change and percent change from baseline in the PP-NRS. The measument will perform via using the peak pruritus-numerical rating scale (PP-NRS) , an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
  The PP-NRS was designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours
Efficacy endpoint will be assessed through collection and analysis of lesion Assessment- (PP-NRS)- responders | up to 7 weeks
  Percent responders in PP-NRS. The measument will perform via using the peak pruritus-numerical rating scale (PP-NRS) , an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
  A responder is defined to have an improvement of at least 4 points on the 11-point PP-NRS scale

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Fachklinik Bad Bentheim - Dermatologische Studienambulanz, Bensheim
  - Rothhaar Studien GmbH, Berlin

IPD SHARING:
Plan to Share IPD: No